CLINICAL TRIAL: NCT03893760
Title: Assessment of Right Ventricular Function in Advanced Heart Failure: Feasibility and Reliability of Right Ventricular Elastance
Brief Title: Assessment of Right Ventricular Function in Advanced Heart Failure
Status: Completed | Type: Observational
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Principal Investigator, ITAB - Institute for Advanced Biomedical Technologies
Other Study IDs: NGCH001
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Dilated Cardiomyopathy; Heart Failure
Keywords: heart Failure; ventricular elastance; dilated cardiomyopathy; right heart systolic function; right ventriculo-arterial coupling
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No Pulonary Hypertension: the presence of mean pulmonary pressures (PAPm) at the right heart catheterization < 25 mmHg
  Interventions: Diagnostic Test: Ventriculo-arterial coupling assessment (R-V/A)
- Postcapillary Pulmonary Hypertension: PAPm ≥ 25 mmHg and postcapillary wedge pressure (PCWP) >15 mmHg
  Interventions: Diagnostic Test: Ventriculo-arterial coupling assessment (R-V/A)
- combined postcapillary/precapillary Pulmonary Hypertension: PAPm ≥ 25 mmHg, PAWP >15 mmHg and diastolic peak gradient (DPG - diastolic pulmonary pressure - PCWP) ≥7 mmHg and/or pulmonary vascular resistence (PVR) >3 WU, where available.
  Interventions: Diagnostic Test: Ventriculo-arterial coupling assessment (R-V/A)

INTERVENTIONS:
Diagnostic Test: Ventriculo-arterial coupling assessment (R-V/A) — R-V/A was achieved by computing the R-Elv/P-Ea ratio (Right ventricular elastance/Pulmonary arterial elastance). R-Elv was computed as PAPm / end-systolic area (ESA) of the right ventricle. P-Ea was obtained as (PAPm-PCWP)/ right ventricle stroke volume (R-SV).

SUMMARY:
We examined the feasibility and reliability of a combined echocardiographic and right heart catheterization (RHC) approach for right ventriculo/arterial (R-V/A) coupling assessment in HF patients with dilated cardiomyopathy (D-CMP).

DETAILED DESCRIPTION:
This is a single center, retrospective cross-sectional study. In 2016-17, for 6 months, we evaluated for eligibility 81 consecutive D-CMP patients afferent to "Niguarda Great Metropolitan Hospital" for RHC and echocardiography. All participants underwent the exams in the context of heart-transplant or advanced HF evaluation. Inclusion criteria were: 18 years old, given informed consent, D-CMP, New York Heart Association (NYHA) functional class II or III and reduced EF (≤ 35%). On the contrary, exclusion criteria were: missing the inclusion criteria and refused informed consent. The final sample consisted of 68 study participants (mean age 64±7 years, 82 % male).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Given informed consent
* D-CMP
* New York Heart Association (NYHA) functional class II or III
* Reduced EF (≤ 35%)

Exclusion Criteria:

* Missing the inclusion criteria
* Refused informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants underwent the exams in the context of heart-transplant or advanced HF evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with altered Right ventriculo/arterial (R-V/A) coupling over PAPm and Pulmonary Hypertension types | up to 24 weeks
  Significant correlations and augmentation over PAPm and Pulmonay Hypertension

SECONDARY OUTCOMES:
Rate of agreement in Right ventriculo/arterial (R-V/A) coupling assessment | up to 24 weeks
  Two independent physicians, both experts in echocardiography, independently re-examined 40 studies, randomly selected from all the acquired echocardiographic images. In order to test the R-V/A coupling interobserver agreement

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bianco, MD, Principal Investigator — Institute of Cardiology - University "G. d'Annunzio" - Chieti, Italy
Locations (2):
- Italy (2):
  - University "G. d'Annunzio", Chieti
  - Niguarda Great Metropolitan Hospital, Milan

IPD SHARING:
Plan to Share IPD: No